CLINICAL TRIAL: NCT02242890
Title: Pilot #2: The Woman-to-Woman Dissemination Project: Harnessing the Power of Social Networks to Increase IUC Use
Brief Title: Pilot #2 of Social Network Intrauterine Contraceptive (IUC) Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: William and Flora Hewlett Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2012-8070-2
Record Dates: First submitted 2014-09-15; First posted 2014-09-17 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-09

CONDITIONS: Attitudes
Keywords: intrauterine contraception (IUC); social networks; social influence; diffusion of innovation; intrauterine device (IUD); LARC
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Contraception Information Packet (Other): Everyone in the study will receive the intervention, which is an information packet designed to facilitate conversations among peers about intrauterine contraception.
  Interventions: Behavioral: Contraception Information Packet

INTERVENTIONS:
Behavioral: Contraception Information Packet — The intervention will consist of brief education about IUC and development of interpersonal skills, including how to initiate conversations about reproductive health issues in social settings and debunking common IUC myths.

SUMMARY:
This study has two goals: 1) to test an approach to helping women who use intrauterine contraception (IUC) spread the word about this type of long-lasting, highly effective birth control method among their friends and family and; 2) to test ways of getting in touch with these women's friends and family so that investigators can track whether this approach is effective at spreading birth control information through social groups.

DETAILED DESCRIPTION:
Pilot of peer IUC intervention:

Investigators will assess the feasibility and acceptability of a low-cost intervention implemented at a clinic providing family planning care. The intervention was first piloted in the an earlier phase of this study (ClincalTrials.gov ID: NCT01965743) which is currently in the analysis phase. Based off of participant feedback from this first pilot, investigators have revised and optimized the intervention which investigators will be testing again here at a new clinic and with a new population.

New IUC users as well as experienced IUC users will be recruited as "dissemination agents" to provide information about the option of IUC to their peers. Ten to sixteen IUC users will be recruited from a family planning clinic to receive the intervention.The intervention which will be delivered by a clinic staff member to new or existing IUC users includes handing her a packet of pamphlets, encouraging her to sign up for a series of SMS messages, and informing her about the intervention's website. The content on the intervention across all media forms consists of a brief education about IUC and development of interpersonal skills for IUC users, including how to initiate conversations about reproductive health issues and their personal experience with IUC in social settings.

Investigators will conduct baseline and 3 month quantitative surveys as well as 3-month qualitative interviews of dissemination agents to asses the feasibility and impact of the intervention on IUC knowledge, attitudes and social communication practices. As described in more detail below, investigators will also enroll the social contacts of dissemination agents to measure the effect of the intervention on their IUC knowledge and attitudes.

At the completion of dissemination agent enrollment and intervention implementation in clinic, investigators will also conduct a focus group with clinic staff about the feasibility of implementing the intervention in the clinical setting.

Test of snowball sampling for social network analysis:

The social contacts of dissemination agents will be recruited via one of two snowball sampling methods: baseline or follow up recruitment methods. Dissemination agents will be randomized into each recruitment arm. In both recruitment arms, dissemination agents will list at baseline and at 3 month follow up their female social contacts between the ages of 15-45 with whom they feel comfortable talking about birth control with.

In the baseline recruitment arm, the dissemination agents within the first 2 weeks of being enrolled will ask their listed social contacts if they are interested in joining a study about birth control and for permission for the dissemination agent to share their contact info with the study staff. Study staff will then reach out to the social contacts whom have shared their contact information with us to ask if they would like to enroll in the study. Social contacts who choose to enroll will complete a baseline survey as well as another follow up survey 3 months from when their respective dissemination agent enrolled.

In the follow up recruitment arm, dissemination agents at 3 months from their enrollment will recruit in the same manner as the baseline arm their social contacts. They will be asked to recruit all social contacts listed at baseline and any additional ones added at 3 months. Social contacts who enroll will complete 1 survey at the time of their enrollment.

In both arms, dissemination agents will receive a small "finder's fee" for each social contact with whom the study is able to make contact with and confirms that she gave the dissemination agent permission to share her contact info.

Investigators will assess which recruitment method is most effective at enrolling members of the dissemination agents' social network and whether social contacts in the baseline arm had more conversations about IUC with their dissemination agents between baseline and follow up due to the presence of recruitment conversations happening concurrently.

A randomly selected sub-set of social contacts in both arms will be selected to complete a more detailed qualitative interview after quantitative data collection is complete. To minimize any potential Hawthorne effect, social contacts will initially be blinded as to the specific aims being assessed, and will be debriefed at the end of the study.

This pilot study will provide the data necessary to prepare for a randomized controlled trial of this intervention.

ELIGIBILITY:
Inclusion Criteria:

Dissemination agents:

* Have an IUD placed for contraception at clinic visit or have existing IUD for contraception
* Speak English
* Age 15-45
* Willing to disclose IUD use to friends and family
* Willing to have research staff contact their friends and family to participate in study related to family planning

Social contacts:

* Age 15-45 Speak English
* Able to get pregnant
* Ever sexually active with men
* Acquainted with dissemination agent
* Makes contact with study team within one month of dissemination agent's enrollment (baseline arm) or within one month of dissemination agent's 3 months follow up (follow up arm)
* Lives in the United States of America.

Clinic staff:

-Able to provide family planning care at clinic where intervention is being implemented.

Exclusion Criteria:

Dissemination agents:

* Using IUD for reason other than contraception
* Unwilling to disclose IUD use to any social contacts
* Unwilling to allow research staff to enroll friends and family in study as social contacts
* Do not speak or understand English

Social contacts:

* Unable to get pregnant
* Do not speak or understand English.

Clinic staff:

-Not working at clinic at time of intervention.

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2015-02; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Acceptability of WhyIUD intervention to intervention participants | 3 months
  Study staff will administer 3-month post-intervention surveys with participants to quantitatively assess their opinions of and engagement with the WhyIUD intervention. Staff will also conduct structured interviews with a selection of participants at 3 months to gather qualitative feedback on the intervention.

SECONDARY OUTCOMES:
Feasability of snowball sampling procedure to obtain social network sample | 3 months
  Study staff will measure the percentage of identified social contacts who participate in the study and their retention during the study period.
Change in IUD-related knowledge among intervention participants | 3 months
  Baseline and 3-month surveys with participants will include measures related to IUD knowledge.
Change in IUD-related attitudes among patient participants | 3 months
  Baseline and 3-month surveys with participants will include measures related to IUD attitudes.
Change in IUD-related social communication among patient participants | 3 months
  Baseline and 3-month surveys with participants will include measures related to social communication with friends and family about the IUD.
Acceptability of WhyIUD intervention to clinic staff | 1 month
  After the 1-month period during which the intervention is actively delivered in clinic, study staff will conduct a focus group with clinic personnel who were involved in the delivery of WhyIUD to assess acceptability by gathering their opinions and experience of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Dehlendorf, MD, MAS, Principal Investigator — University of California, San Francisco
Locations (1):
- Planned Parenthood North Highlands, North Highlands, California, United States